CLINICAL TRIAL: NCT06209892
Title: Prolonged Anticoagulation Therapy on the Prognosis of Patients With Left Ventricular
Brief Title: Prolonged Anticoagulation Therapy on the Prognosis of Patients With Left Ventricular Thrombosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Weihua Song, MD, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJHPA-2023-017-014
Record Dates: First submitted 2024-01-06; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Embolism and Thrombosis; Anticoagulation
MeSH Terms: conditions — Embolism and Thrombosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional anticoagulation group (No Intervention)
- Extended anticoagulation group (Experimental)
  Interventions: Procedure: Extended anticoagulation

INTERVENTIONS:
Procedure: Extended anticoagulation — This study plan will extend the duration of rivaroxaban 20mg in the experimental group to 12 months. The regular anticoagulation group will take the drug for 6 months
  Arms: Extended anticoagulation group

SUMMARY:
A single-center, open-label, exploratory randomized controlled study is proposed with the following objectives: whether prolonging the duration of anticoagulation to 12 months, compared with 6 months of routine anticoagulation, helps to reduce major adverse cardiovascular and cerebrovascular events in patients with left ventricular thrombosis and to reduce recurrence of thrombosis, as well as to assess their bleeding risk.

Patients with a definite diagnosis of left ventricular thrombus and age ≥18 years were included in cardiac ultrasound (including general ultrasound and sonography) and other examinations during hospitalization and outpatient visits. Exclusion criteria were detailed in the study protocol.

GROUPING: According to the duration of anticoagulation, they were divided into extended anticoagulation group (12 months) and conventional anticoagulation group (6 months).

INTERVENTION: This study is planned to extend the administration of rivaroxaban (Pulsatilla) 20 mg to 12 months in the experimental group. The conventional anticoagulation group will take the drug for 6 months Study Endpoints: The primary efficacy endpoint is a major cardiovascular-vascular adverse event at 1 year; the primary safety endpoint is bleeding of grade 3 or higher as defined by the BARC classification at 1 year.

Patient Follow-up Program: Subjects will require a total of 12 on-site follow-up visits (one per month) for safety evaluation, efficacy evaluation, medication adherence evaluation, and imaging follow-up at months 3, 6, and 12.

ELIGIBILITY:
Inclusion Criteria:

①Patients who have been clearly diagnosed with left ventricular thrombus by inpatient or outpatient cardiac ultrasound (including general ultrasound and acoustic imaging).

②Age >= 18 years old

Exclusion Criteria:

* Patients do not agree to participate in the study or have poor compliance in the past

  * Contraindication to anticoagulation or allergy to anticoagulants ③Have received oral anticoagulation after diagnosis of left ventricular thrombus.

    * Have undergone or are planning to undergo surgical procedures including left ventricular appendage thrombectomy, heart transplantation, ventricular wall tumor collapse, or valve replacement.

      * Presence of other long-term indications for anticoagulation, such as mechanical valve implantation, atrial fibrillation, etc.

        * Requirement for treatment with Tegretol and inability to change to clopidogrel bisulfate ⑦Presence of known malignant tumors, severe hepatic dysfunction (Child-Pugh classification B or less), severe renal dysfunction (creatinine clearance <30ml/min), anemia (Hb <100g/L), coagulation disorders and other underlying diseases, or life expectancy <3 years ⑧ Female patients are pregnant or breastfeeding ⑨ Patients with antiphospholipid syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoint | Patient completes one year of follow-up
  for major cardiovascular and cerebrovascular adverse events at 1 year, including: all-cause mortality, nonfatal heart attack, ischemic stroke, and acute peripheral artery embolism. fatal heart attack, ischemic stroke, and acute peripheral artery embolism

SECONDARY OUTCOMES:
secondary endpoint | Patient during one year of follow-up
  Dissolution of left ventricular thrombus confirmed by cardiac ultrasound and no recurrence detected and/or recurrence of left ventricular thrombus detected by cardiac ultrasound after dissolution of left ventricular thrombus

OTHER OUTCOMES:
Primary safety endpoint | Patient during one year of follow-up
  Bleeding of grade 3 or higher as defined by the BARC classification at 1 year

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bulluck H, Vincent M, Hausenloy DJ. Optimizing the Detection of Left Ventricular Thrombus Following Acute Myocardial Infarction in the Current Era. JAMA Cardiol. 2018 Nov 1;3(11):1128-1129. doi: 10.1001/jamacardio.2018.3136. No abstract available. PMID 30285032
- [Result] Maniwa N, Fujino M, Nakai M, Nishimura K, Miyamoto Y, Kataoka Y, Asaumi Y, Tahara Y, Nakanishi M, Anzai T, Kusano K, Akasaka T, Goto Y, Noguchi T, Yasuda S. Anticoagulation combined with antiplatelet therapy in patients with left ventricular thrombus after first acute myocardial infarction. Eur Heart J. 2018 Jan 14;39(3):201-208. doi: 10.1093/eurheartj/ehx551. PMID 29029233
- [Result] Lattuca B, Bouziri N, Kerneis M, Portal JJ, Zhou J, Hauguel-Moreau M, Mameri A, Zeitouni M, Guedeney P, Hammoudi N, Isnard R, Pousset F, Collet JP, Vicaut E, Montalescot G, Silvain J; ACTION Study Group. Antithrombotic Therapy for Patients With Left Ventricular Mural Thrombus. J Am Coll Cardiol. 2020 Apr 14;75(14):1676-1685. doi: 10.1016/j.jacc.2020.01.057. PMID 32273033